CLINICAL TRIAL: NCT06729463
Title: IKBKB Gene Polymorphism (Single Nucleotide Polymorphism) (SNP) in Psoriatic and Psoriatic Arthritis Patients and Its Relation With Response to Systemic Biologic Therapy
Brief Title: IKBKB Gene Polymorphism (Single Nucleotide Polymorphism) (SNP) in Psoriatic and Psoriatic Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Fatma Abdel-monem Mahmoud, Resident of Dermatology, Venereology and Andrology., South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fatma Abdel-Monem
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Adalimumab; secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Humira Group (Active Comparator): About 20 patients suffering from psoriasis disease and they will take Humira vials about 40 mg every two weeks by subcutaneous injection for 3 months
  Interventions: Drug: Humira
- Group B: Cosentyx Group (Active Comparator): About 20 patients suffering from severe psoriasis will take Cosentyx vials by intravenous infusion as :
  1-Loading dose about(300 mg) then decreasing the dose to be 150 mg every month for 3 months.
  Interventions: Drug: Humira
- Group C: control Group (Placebo Comparator): About 10 Healthy participants and will take no medical treatment
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: Humira — Assess the pharmacogenetic association between IKBKB gene polymorphism (SNPs) in psoriatic patients taking systemic biologic therapy
  Other Names: Cosentyx

SUMMARY:
Psoriasis is a chronic inflammatory skin disease characterized by scaly indurated erythema. It impairs patients' quality of life enormously.

Psoriasis refers to a persistent inflammatory illness of the skin and joints. It also impacts roughly 2%-3% of the inhabitants of the universe

DETAILED DESCRIPTION:
The exact aetiopathogenesis of psoriasis is not completely explained. Pathological mechanism involves skin inflammation and hyperproliferation of keratinocytes induced innate and adaptive immune cells. Genetic, immunological and environmental factors are considered the most important aetiologies.

Psoriatic arthritis, which is characterized by dactylitis and enthesis, is closely associated with psoriasis. Up to 30-40% of patients with psoriasis will develop PsA, with an average of 10 years between psoriasis and PsA . The overlapping of genetic variations and inflammatory mediators involved in psoriasis and PsA implies a common pathogenic mechanism between the two diseases.

Psoriasis is a chronic relapsing disease, which often necessitates a long-term therapy. Mild to moderate psoriasis can be treated topically with a combination of glucocorticoids, vitamin D analogues, and phototherapy. Moderate to severe psoriasis often requires systemic treatment. The presence of comorbidities such as psoriasis arthritis is also highly relevant in treatment selection.

Oral treatments include traditional agents such as methotrexate, acitretin, cyclosporine, and the advanced small molecule apremilast, which is a phosphodiesterase 4 inhibitor. Oral treatments include traditional agents such as methotrexate, acitretin, cyclosporine, and the advanced small molecule apremilast, which is a phosphodiesterase 4 inhibitor.

The American Academy of Dermatology-National Psoriasis Foundation guidelines recommend biologics as an option for first-line treatment of moderate to severe plaque psoriasis because of their efficacy in treating it and acceptable safety profiles.

Specifically, inhibitors to tumour necrosis factor α (TNF-α) include etanercept, adalimumab, certolizumab, and infliximab. Other biologics inhibit cytokines such as the p40 subunit of the cytokines IL-12 and IL-13 (ustekinumab), IL-17 (secukinumab, ixekizumab, bimekizumab, and brodalumab), and the p19 subunit of IL-23 (guselkumab, tildrakizumab, risankizumab, and mirikizumab). Biologics that inhibit TNF-α, p40IL-12/23, and IL-17 are also approved for the treatment of psoriatic arthritis.

The NF-κB pathway would play an important role in psoriasis. In this way, the NF-κB is regarded as a mediator between immunity and the keratinocyte alteration characteristic of psoriasis .

This role is also supported by the fact that the blockade of the NF-κB binding sites would reduce the expression of several proinflammatory cytokines implicated in psoriasis. The transcriptional activity of NF-κB is regulated by several cytoplasmic inhibitors. Among these nuclear inhibitors, IκBKB (encoded by NFKBIZ) would play a prominent role in the pathogenesis of psoriasis.

IκBKB(Inhibitor of nuclear factor-kappa B subunit ζ ) is induced by several proinflammatory molecules. In particular, its expression is regulated by IL-17A and might contribute to the activation of Th17-mediated pathways. Therefore, IκBζ( IκBKB) plays an important role in the pathogenesis of psoriatic disease through IL-17-mediated mechanisms.

Recently, genome-wide association studies (GWAS) have found a significant association between psoriasis and single-nucleotide polymorphisms (SNPs) within NFKB1, NFKBIA, and NFKBIZ

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 16 and 60 years proved having psoriasis diagnosed clinically for at least 6 months and who have a severity grade of moderate to severe, defined as a Psoriasis Area and Severity Index (PASI) score greater than 10, and involvement of greater than 10% of the body surface area (BSA) with or without psoriatic arthritis

Exclusion Criteria:

* Patient receiving immune suppressive drugs.
* Patients having malignancy.
* Pregnant or lactating female.
* Patients having liver disease ( Hepatitis)
* Patients having comorbid and/or uncontrolled renal, cardiac, vascular, and hepatic diseases or symptoms.
* Active infection or human immunodeficiency virus (HIV)
* Tuberculosis

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Treatment of the Psoriasis disease | 3 months
  Evaluation the clinical efficacy of biological therapy in patients of psoriasis and assessing the relation between the drug response and IKBKB mutation

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Professor, Study Chair — Dermatology, Venereology, and Andrology Department, Faculty of Medicine, South Valley University, Egypt
Locations (1):
- South Valley Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided